CLINICAL TRIAL: NCT04256993
Title: Rates of Bone Fractures and Survival in Metastatic Castration-resistant PRostate Cancer (mCRPC) PatiEnts Treated With Radium 223 in Routine Clinical practIce in SwedEn
Brief Title: PRECISE, a Study to Gather More Information About Bone Fractures and Survival in Castration-resistant PRostate Cancer (CRPC) patiEnts Treated With Radium-223 in Routine Clinical practIce in SwedEn
Acronym: PRECISE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20437
Record Dates: First submitted 2020-02-04; First posted 2020-02-05 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Prostate cancer metastatic; Prostate cancer; Bone fractures; Overall survival
MeSH Terms: conditions — Prostatic Neoplasms; Fractures, Bone | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ra-223 initiators: Patients diagnosed with mCRPC (Metastatic Castration-Resistant Prostate Cancer) who start treatment with Ra-223. Patients will be identified from the "Patient-overview Prostate Cancer" (PPC), a sub-registry of the Prostate Cancer data Base Sweden (PCBaSe) data set.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)
- Initiators of other standard of care: The comparator cohort will be patients using standard of care other than Ra-223.
  Interventions: Drug: Other standard care

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Follow the physician's prescription in routine clinical practice. This study does not involve prescription of the drugs.
  Groups: Ra-223 initiators
Drug: Other standard care — Docetaxel, cabazitaxel, enzalutamide, abiraterone and others standard of care following the physician's prescription in routine clinical practice.
  Groups: Initiators of other standard of care

SUMMARY:
In this observational study researchers want to gather more information about bone fractures and survival in castration-resistant prostate cancer (CRPC) patients treated with radium-223 in routine clinical practice in Sweden. The goal is to estimate the proportion of new cases (incidence) of symptomatic bone fractures and to estimate the proportion of death occurred in years of observation time per person (person years). Radium-223 (Ra-223) is an alpha particle-emitting radioactive agent approved for the treatment of men with metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate, i.e., the patient is registered in the NPCR (histology other than adenocarcinomas are not registered in the NPCR).
* Start of Ra-223 treatment for mCRPC as an n-th line of treatment, where "n" goes from 1 to 4.
* ECOG performance status of 0-2 at treatment initiation. We will assume that patients starting any of the systemic therapies under study have a performance status of 0-2.

Exclusion Criteria:

* Prior use of Ra-223
* Patients that have participated in a Ra-223 RCT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises men with mCRPC in the PPC (Patient-overview Prostate Cancer) PCBaSe data set during the study time frame, with the potential addition of men with mCRPC in the Karolinska Institutet data sets.
Sampling Method: Non-Probability Sample
Enrollment: 1434 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Bone fractures requiring admission to a hospital or treated in an outpatient setting, as recorded or captured in the PCBaSe | Retrospectively analysis from November 2013 to December 2018
  PCBaSe: Prostate Cancer data Base Sweden

SECONDARY OUTCOMES:
Death due to all causes | Retrospectively analysis from November 2013 to December 2018
Death due to prostate cancer | Retrospectively analysis from November 2013 to December 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Database Study, Database Study, Sweden

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/